CLINICAL TRIAL: NCT05152355
Title: Multi-center, Single Blind, Randomized, Parallel Study to Compare the Clinical Efficacy and Safety of Dusama (Budesonide) HFA MDI With Pulmicort (Budesonide) Turbuhaler in Mild to Moderate Chinese Asthma Patients
Brief Title: Clinical Equivalence of Budesonide HFA MDI Versus Budesonide Turbuhaler in Mild to Moderate Chinese Asthma Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Intech Biopharm Ltd. (Industry)
Collaborators: GCP ClinPlus Co., Ltd. (Unknown); Beijing Aicomer Pharmaceutical Technology Co., Ltd. (Unknown); Key Tech (Unknown); Healthcare Inc (Unknown); Peking University People's Hospital (Other); Beijing Friendship Hospital (Other); Tianjin First Central Hospital (Other); Bao Gang Hospital (Unknown); The Affiliated Hospital of Inner Mongolia Medical University (Other); Beijing Yi Hua Hospital Management Co., Ltd (Unknown); The Second Hospital of Hebei Medical University (Other); The First Affiliated Hospital of Shanxi Medical University (Other); Shaanxi Provincial People's Hospital (Other); Jining Medical University (Other); Qingdao Municipal Hospital (Other); Daqing Oil Field Hospital (Other); First Affiliated Hospital of Jinan University (Other); Meizhou People's Hospital (Other); Meiheko Central Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INTB011H01
Record Dates: First submitted 2020-07-30; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-08

CONDITIONS: Asthma
Keywords: budesonide; MDI; DPI; China; Asthma
MeSH Terms: conditions — Asthma | interventions — Nebulizers and Vaporizers; Inhalation; Budesonide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Budesonide HFA MDI (Treatment A) (Experimental): Participants assigned to Experimental arm will inhaled 2 puffs of budesonide 200 mcg HFA MDI bid (am 08:00 and pm 16:00) for 4 weeks
  Interventions: Drug: Budesonide 200 microgram/Puff, HFA MDI
- Budesonide DPI (Turbuhaler) (Treatment B) (Active Comparator): Participants assigned to Active Comparator arm will inhaled 4 puffs of budesonide 100 mcg powder for inhalation bid (am 08:00 and pm 16:00) for 4 weeks
  Interventions: Drug: Budesonide 100 microgram/Actuation Powder for Inhalation

INTERVENTIONS:
Drug: Budesonide 200 microgram/Puff, HFA MDI — Participants will inhaled 2 puffs of budesonide 200 mcg HFA MDI bid (am 08:00 and pm 16:00) for 4 weeks, if necessary rescue Ventolin (Salbutamol Sulfate) 100 mcg 2 puffs could be used with maximum daily dose of 8 puffs.
  Other Names: Duasma 200 mcg inhaler
  Arms: Budesonide HFA MDI (Treatment A)
Drug: Budesonide 100 microgram/Actuation Powder for Inhalation — Participants will inhaled 4 puffs of budesonide 100 mcg DPI bid (am 08:00 and pm 16:00) for 4 weeks, if necessary rescue Ventolin (Salbutamol Sulfate) 100 mcg 2 puffs could be used with maximum daily dose of 8 puffs.
  Other Names: Pulmicort 100 mcg Turbuhaler
  Arms: Budesonide DPI (Turbuhaler) (Treatment B)

SUMMARY:
The primary objective of this study is to compare the efficacy and safety of budesonide HFA MDI 200 mcg 2 puffs BID versus budesonide DPI (Turbuhaler) 100 mcg 4 puffs BID in Chinese mild to moderate Asthma patients.

DETAILED DESCRIPTION:
A total of 270 Chinese mild to moderate Asthma patients will be enrolled and 230 will be completed in this multi-center, randomized, single blind, parallel efficacy and safety comparison study of budesonide HFA MDI 200 mcg 2 puffs BID versus budesonide DPI (Turbuhaler) 100 mcg 4 puffs BID.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 70 years old and diagnosed as Asthma in clinics
* Diagnosed as Asthma according to the 2016 Asthma guidance of Chinese Thoracic Society, and without administer corticosteroids within three months, either new or old patients
* FEV1 predicted ≧ 60%
* Patients is willing to participate the study and signed the Informed Consent Form

Exclusion Criteria:

* Allergy to budesonide or salbutamol
* Infections of Respiratory tract, nasal-sinus and ear within 4 weeks before enrollment
* Severe nasal allergy and need the treatment of corticostreoids and histamines.
* Severe cardiovascular disease history
* Has used leukotriene receptor antagonist (Montelukast, Pranlukast, Zafirlukast etc.) within 2 weeks before enrollment
* Severe cognition or mental disorder and can not cooperation with the treatment
* Significant liver dysfunction, AST, ALT > 3 X normal upper limits, CR > 1.5 X normal upper limits
* Patients with uncontrolled diabetes or fasting blood glucose > 10 mmol/L
* Patients currently receiving beta-antagonists or beta-agonists treatment (including eye drops)
* Patients who has contraindications to beta2-agonists
* Patients who has participated others drug's clinical study within three months
* Female patients who are pregnant or lactation or prepare to pregnant
* Any conditions which the investigators considered not suitable to enrolled

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2021-05-09 (Actual); Study Completion 2021-05-09 (Actual)

PRIMARY OUTCOMES:
Change from base line of FEV1 | Week 0, 2 and 4
  The change from base line of forced expiratory volume in one second after 4 weeks treatment

SECONDARY OUTCOMES:
Mean change from base line of morning and evening PEF | Week 0 and 4
  The mean change from base line of morning and evening PEF (peak expiratory flow)
Change from base line of FVC | Week 0 and 4
  The changes from base line of FVC after 4 weeks treatment
Change from base line of FEV1/FVC ratio | Week 0 and 4
  The changes from base line of FEV1/FVC ratio after 4 weeks treatment
Change from base line of FEF25% | Week 0 and 4
  The changes from base line of FEF25% after 4 weeks treatment
Change from base line of FEF50% | Week 0 and 4
  The changes from base line of FEF50% after 4 weeks treatment
Change from base line of FEF75% | Week 0 and 4
  The changes from base line of FEF75% after 4 weeks treatment
Change from base line of ACT | Week 0, 2 and 4
  The change from base line of Asthma Control Test after 4 weeks treatment
Daily PEF variability | during week 0 to 4
  The Daily PEF variability (= (daily highest PEF-daily lowest PEF)X2/((daily highest PEF+daily lowest PEF) X 100% during the whole treatment period
Weekly PEF variability | during week 0 to 4
  The Weekly PEF variability (= (biweely highest PEF-biweekly lowest PEF)X2/((biweekly highest PEF+biweekly lowest PEF) X 100% during the whole treatment period
Changes of day time and night time symptom | during week 0 to 4
  The changes of day time and night time symptom during the treatment period
Subjects number with acute exacerbation | during week 0 to 4
  The total number of subjects with acute exacerbation during treatment period
Total amount of rescue medication, Ventolin 100 mcg inhaler, used | during week 0 to 4
  The total amount of doses of rescue medication, Ventolin 100 mcg inhaler, used during the treatment period
Percentage of days without symptom | during week 0 to 4
  The percentage of days without asthma symptom during the treatment period
Percentage of days without using rescue medicine | during week 0 to 4
  The percentage of days without using rescue medicine during the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Wei Hsiu Wu, MBA, Study Chair — Intech Biopharm
Locations (13):
- China (13):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - Meizhou People's Hospital, Meizhou, Guangdong
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Daqing Oil Field Hospital, Daqing, Heilongjiang
  - Bao Gang Hospital, Baotou, Inner Mongolia
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Meiheko Central Hospital, Tonghua, Jilin
  - Affiliated Hospital of Jining Medical University, Jining, Shandon
  - QingDao Municipal Hospital, Qingdao, Shandon
  - The First Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - Tianjin First Central Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No